CLINICAL TRIAL: NCT01552096
Title: A Comparative Study of the Effects of Pre-incisional Infiltration of Tramadol or Lidocaine on the Inflammatory Response After Tonsillectomy.
Brief Title: Tramadol Versus Lidocaine Infiltration for Tonsillectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #2012082
Record Dates: First submitted 2012-03-05; First posted 2012-03-13 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Peri-tonsillar Analgesic Infiltration; Tonsillectomy; Postoperative Pain; Inflammatory Response
Keywords: Anaesthesia; tonsillectomy; inflammatory response; stress response; tramadol; lidocaine
MeSH Terms: conditions — Pain, Postoperative; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): The placebo group (n=30) will receive a submucosal infiltration with 3 mL of normal saline (1.5 ml around each tonsil), 3 minutes before surgical incision.
  Interventions: Drug: peritonsillar infiltration
- lidocaine (Active Comparator): will receive a total of 2 mg.kg-1 of 2% lidocaine HCl (Xylocaine, Astra-Zeneca,) in 3 mL of normal saline (1.5 ml around each tonsil), 5 minutes before surgical incision.
  Interventions: Drug: peritonsillar infiltration
- Tramadol (Experimental): (n=30) will receive a submucosal infiltration with 2 mg kg-1 tramadol in 3 mL of normal saline (1.5 ml around each tonsil), 3 minutes before surgical incision.
  Interventions: Drug: peritonsillar infiltration

INTERVENTIONS:
Drug: peritonsillar infiltration — 1.5 ml around each tonsil, 3 minutes before surgical incision as per group description
  Other Names: as in description

SUMMARY:
The investigators postulate that the use of pre-incisional peritonsillar infiltration of tramadol or lidocaine reduces both the inflammatory response and postoperative analgesic consumption, without harmful effects. Therefore, the present study is designed to evaluate the effects of infiltration of tramadol or lidocaine on the postoperative acute-phase serum protein, C-reactive protein, and analgesic consumption after tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II preschool children aged 2-6 years, undergoing elective tonsillectomy with or without adenoidectomy, under general anaesthesia. Indications for tonsillectomy will be chronic recurrent tonsillitis or tonsillar hypertrophy

Exclusion Criteria:

* Patients with a history of allergy to tramadol or amide local anaesthetics, epilepsy, or taking cardiovascular, antihypertensive, steroids, or anti-inflammatory medications, those with cardiac, liver, or kidney diseases, or any underlying systemic diseases or acute infectious processes will be excluded from the study. All operations will be performed, using an electro-dissection technique, by the same surgeon.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
inflammatory and stress response | 24 hours
  CRP Acute phase protein

SECONDARY OUTCOMES:
Hemodynamic changes | 24 hours
  MBP HR
pain score | 24 hours
  VAS The time to first request for analgesia and the number of subjects receiving meperidine during the first 12 hours will be recorded.
Side-effects | 24 hours
  postoperative stridor, laryngospasm, cyanosis, bleeding, seizures, sedation (four-point verbal rating scores (VRS): awake, drowsy, rousable or deep sleep); nausea and vomiting (0: no nausea; 1: nausea no vomiting; 2: nausea and vomiting), respiratory depression (ventilatory frequency 10), and desaturation (92%), at 0, 1, 2, 4, 6, 8, and 12 h after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: laila Telmesani, MD, Principal Investigator — UD; Hany A. Mowafi, MD, Study Chair — Associate Professor; Alaa M. Khidr, MD, Study Chair — Assistant Consultant; Abdulhadi Al'Saflan, MD, Study Chair — Assistant Consultant
Locations (2):
- Saudi Arabia (2):
  - Dammam University KFHU, Khobar, EP
  - UD-KFHU, Khobar, EP